CLINICAL TRIAL: NCT03757390
Title: An Open-label, Randomized, Single-dose Crossover Study to Evaluate the Pharmacokinetics, Safety and Tolerability of CJ-30060 in Healthy Subjects
Brief Title: Bioequivalence Study of CJ-30060 in Healthy Volunteers
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: HK inno.N Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CJ_EXR_104
Record Dates: First submitted 2018-11-25; First posted 2018-11-28 (Actual); Last update posted 2018-11-28 (Actual); Status verified 2018-11

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — Amlodipine, Valsartan Drug Combination; Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence 1 (Experimental): * period 1: receive Exforge® tab 5/160mg, Crestor® tab 10mg
  * period 2: receive CJ-30060 5/160/10mg
  Interventions: Drug: Exforge® tab 5/160mg, Crestor® tab 10mg; Drug: CJ-30060 5/160/10mg
- Sequence 2 (Experimental): * period 1: receive CJ-30060 5/160/10mg
  * period 2: receive Exforge® tab 5/160mg, Crestor® tab 10mg
  Interventions: Drug: Exforge® tab 5/160mg, Crestor® tab 10mg; Drug: CJ-30060 5/160/10mg

INTERVENTIONS:
Drug: Exforge® tab 5/160mg, Crestor® tab 10mg — co-administration of Amlodipine 5mg/Valsartan 160mg(combination drug) and Rosuvastation 10mg
Drug: CJ-30060 5/160/10mg — Fixed-dose combination drug containing Amlodipine 5mg and Valsartan 160mg and Rosuvastatin 10mg

SUMMARY:
To compare the pharmacokinetics and safety after a single dose administration of CJ-30060 and Exforge® 5/160mg, Crestor® 10mg in healthy volunteers.

DETAILED DESCRIPTION:
The purpose of this study is to compare the pharmacokinetics and safety after a single dose administration of CJ-30060 and Exforge® 5/160mg, Crestor® 10mg in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers aged 20 to 45 years at screening
* BMI: 18~29.9kg/㎡
* Body weight ≥50kg
* Subjects who decided to participate in the study and signed informed consent form voluntarily after receiving detailed explanation of the study and fully understanding

Exclusion Criteria:

* Subjects who had a medical history of severe cardiovascular, respiratory, hepatobiliary, renal, hematological, gastrointestinal, endocrinological, immunological, dermatological or neuropsychological disease
* Subjects who have symptoms of an acute disease within 28days before first administration
* Subjects who have clinically significant active, chronic disease
* Subjects who fall under the criteria below in laboratory test

  * AST/ALT > UNL (upper normal limit) × 2
  * Total bilirubin > UNL × 1.5
  * CrCL < 50mL/min
  * CPK > UNL × 2.5
* Subjects with clinically significant low blood pressure at screening test(systolic blood presure is less than 100mmHg or diastolic blood pressure is less than 60mmHg)
* Subjects with any positive reaction in HBsAg, anti-HCV Ab, anti HIV Ab, VDRL tests

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Estimated)
Dates: Start 2018-11-09 (Actual); Primary Completion 2018-12-14 (Estimated); Study Completion 2018-12-14 (Estimated)

PRIMARY OUTCOMES:
Cmax of amlodipine | Up to 144 hours post-dose
Cmax of valsartan | Up to 48 hours post-dose
Cmax of rosuvastatin | Up to 72 hours post-dose
AUClast of amlodipine | Up to 144 hours post-dose
AUClast of valsartan | Up to 48 hours post-dose
AUClast of rosuvastatin | Up to 72 hours post-dose

SECONDARY OUTCOMES:
AUCinf of amlodipine, valsartan, rosuvastatin | Up to 144 hours post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Ji Young Park, PhD, Principal Investigator — Korea University Anam Hospital
Locations (1):
- Korea University Anam Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No